CLINICAL TRIAL: NCT03341065
Title: Comparisons of Two Types of Robot Assisted Gait Training: Exoskeleton Type Robot vs. End-effector Type Robot: Randomized Controlled Trial
Brief Title: Comparisons of Two Types of Robot Assisted Gait Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Principal Investigator, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRC-2016-01-006
Record Dates: First submitted 2017-10-22; First posted 2017-11-14 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Stroke; Robot Assisted Gait Training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- exoskeleton type robot (Experimental): exoskeleton type robot assisted gait training (Lokomat orthosis)
  Interventions: Device: exoskeleton type robot
- end-effector type robot (Experimental): end-effector type robot assisted gait training (G-EO system)
  Interventions: Device: end-effector type robot

INTERVENTIONS:
Device: exoskeleton type robot
  Arms: exoskeleton type robot
Device: end-effector type robot
  Arms: end-effector type robot

SUMMARY:
Comparisons of Two Types of Robot Assisted Gait Training: Exoskeleton Type Robot vs. End-effector Type Robot: Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Ankle dorsiflexor strength: medical research council scale 2 or 3
* Functional ambulation category score 3

Exclusion Criteria:

* History of surgery of affected lower limb
* Fracture of affected lower limb

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of Range of motion of ankle joint at 4 weeks | 4 weeks from baseline
  ankle joint motion of sagittal plane during gait

SECONDARY OUTCOMES:
Trunk impairment scale | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Trunk impairment scale performs to evaluate the sitting balance and trunk control ability examining static sitting balance, dynamic sitting balance, and coordination, and the maximum score on the subscales are 7, 10, and 6 points, repectively. The total score ranges from 0 to 23 points, a higher score indicating a better trunk performance.
Berg Balance Scale | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Berg Balance Scale assess the functional balance ability of participants with observation of 14 tasks, representing functional movements common in daily life. Each task is scored on a five-point scale (0-4) floolwing the guidelines of the test develpers, and the maximum score on this test is 56 which indicates balance ability within the normal range.
10m walk test | Baseline, 4 weeks from baseline, 8 weeks from baseline
  10m walk test is used to examine gait speed, in which participant was asked to walk on a 14 meter of walkway wearing harness with two conditions; with the fastest speed or with self-selected comfortable speed.
Fugl-Meyer Assessment | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Fugl-Meyer Assessment uses to examine the motor function and coordination of affected lower extremity. It includes 17 items of a 3-point ordinal scale, ranging 0-34, with higher scores indicating lower impairment.
Korean version of Falls efficacy scale | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Korean version of Falls efficacy scale asks subjects to rank their confidence about their ability not to fall while performing a variety of activities of daily living with a maximum score of 100
Range of motion of hip joint | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Hip joint motion of sagittal plane during gait
Range of motion of knee joint | Baseline, 4 weeks from baseline, 8 weeks from baseline
  knee joint motion of sagittal plane during gait
Range of motion of ankle joint | Baseline, 8 weeks from baseline
  ankle joint motion of sagittal plane during gait
Electromyography of lower extremities | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Muscle activity of tibialis anterior, medial gastrocnemius, vastus medialis, biceps femoris, gluteus medius during gait.
Plantar pressure | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Plantar pressure (great toe, little toe, medial meta, lateral meta, medial arch, lateral arch, heel) during gait
Step length, time | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Step length, stance time, swing time, and stride time during gait
Functional Ambulation Category | Baseline, 4 weeks from baseline, 8 weeks from baseline
  Functional Ambulation Category is used to assess gait ability with 6 levels ranging from 0 to 5 on the basis of the amount of physical support required, regardless of use of an assistive device

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Site of the present study — http://nrc.go.kr